CLINICAL TRIAL: NCT03041259
Title: A Phase I/IIa Dose-Escalation Study Evaluating the Safety, Tolerability and Efficacy of Rejuveinix in Combination With Standard Interventional Therapy for Critical Limb Ischemia Patients
Brief Title: Revascularization of Stenosed Vessels Using Optimized Treatment of Rejuveinix for Reversing Endothelial Dysfunction
Acronym: RESTORE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Reven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RPI001
Record Dates: First submitted 2017-01-27; First posted 2017-02-02 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — ascorbic acid, magnesium sulfate heptahydrate, cyanocobalamin, thiamine hydrochloride, riboflavin 5' phosphate, niacinamide, pyridoxine hydrochloride, and calcium D-pantothenate drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rejuveinix Low Dose (Experimental): Intravenous dosing of two doses per week of Rejuveinix
  Interventions: Drug: Rejuveinix Low Dose
- Rejuveinix High Dose (Experimental): Intravenous dosing of two doses per week of Rejuveinix
  Interventions: Drug: Rejuveinix High Dose

INTERVENTIONS:
Drug: Rejuveinix Low Dose — A intravenous administration of Rejuveinix after standard mechanical intervention of blocked peripheral artery
  Other Names: RJX Low
  Arms: Rejuveinix Low Dose
Drug: Rejuveinix High Dose — A intravenous administration of Rejuveinix after standard mechanical intervention of blocked peripheral artery
  Other Names: RJX High
  Arms: Rejuveinix High Dose

SUMMARY:
A Phase I/IIa Dose-Escalation Study Evaluating the Safety, Tolerability and Efficacy of Rejuveinix in Combination With Standard Interventional Therapy for Critical Limb Ischemia Patients with Rutherford Class 4, 5 and 6 Disease

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, multi-center study, comparing MAE and WIQ rates to historical controls to evaluate the safety and efficacy of Rejuveinix for the treatment of patients presenting with symptoms as defined by Rutherford categories 4, 5, or 6, and who have undergone a successful infrainguinal percutaneous intervention within the femoral, femoral-popliteal, popliteal, peroneal, and/or tibial arteries. Treatment at or below the ankle will be permitted (e.g. pedal arteries). This intervention must be successful as defined by ≤ 30% stenosis as determined by angiographic or duplex ultrasound.

Preclinical studies support that Rejuveinix has acute perfusion properties that have the potential to provide synergistic benefits to patients after undergoing current standard of care interventional procedures.

Following an endovascular intervention, in one or more target vessels/lesions, using FDA cleared technology, such as a bare metal stent, angioplasty, and/or atherectomy, patients will receive Rejuveinix as an adjunct therapy. Enrolled subjects will be assigned randomly to one of two groups. Group A will receive two 20 mL treatments of Rejuveinix per week plus one placebo treatment per week comprised of 20 mL 0.9% saline. A dye will be added to the placebo; the dye will be selected from one found in the Orange Book. Group B will receive three treatments of Rejuveinix per week. Each 20 mL treatments will be combined with 100 mL 0.9% saline and administered via intravenous (IV) injection over the course of a minimum of 30 minutes. The study trial will occur for 12 one-week cycles with a washout period of two days between each cycle (a one-week cycle will include either 2 or 3 Rejuveinix treatments depending on the randomized group). Reven will also assess results calculated on four 21-day cycles to allow for a direct comparison to preclinical results.

The goal of the study is to demonstrate Rejuveinix treatment as an adjunctive therapy is non-inferior to historical controls in terms of patient safety, as measured by MAE rates, and efficacy, as assessed by the modified WIQ.

ELIGIBILITY:
Clinical Inclusion Criteria

1. Subject age > 18 and < 90 years of age.
2. Subject has been informed of the nature of the study, agrees to participate and has signed an approved consent form.
3. Subject understands the duration of the study, agrees to follow-up visits and the required testing.
4. Subject has symptomatic lower extremity claudication (meets Rutherford category 4, 5, or 6).
5. Subject has resting ankle-brachial index (ABI) < 0.5, toe pressure <50 mmHg, and/or other evidence suggesting severe PAD (ischemic ulceration, for example).

Anatomic Inclusion Criteria

1. No more than one-week post revascularization, defined as one of the following: PTA, Stent, or Atherectomy.
2. Stenosis in the femoral, femoral-popliteal, popliteal, peroneal, tibial and/or pedal arteries.
3. Angiographic or duplex ultrasound evidence of significant stenosis ≥ 50% DS of target lesion.
4. Target treatment length from 1 to 25 cm (To include single or multifocal lesions within the target lesion segment.
5. Reference vessel diameter (RVD) ≥ 3.5 mm and ≤ 7 mm.
6. Not expected to require further interventional standard of care treatment during study participation (approximately 174 days).

Miscellaneous Inclusion Criteria

1. Anticipated life expectancy >1 year.
2. Has adequate hepatic function defined as total bilirubin < 1.5 mg/dL, serum albumin > 3.0 gm/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 × upper limit of normal (ULN) or < 5 x ULN for subjects with known hepatic metastases.
3. Has adequate renal function defined as serum creatinine < 2.5 × ULN.
4. Has adequate bone marrow function defined as a hemoglobin ≥ 10 mg/dL, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, and platelet count ≥ 100 × 109/L.
5. Must be willing and able to comply with study visits and procedures.
6. Women of childbearing potential (WOCP) must not be pregnant (confirmed by a negative urine pregnancy test prior to enrollment in the trial) nor breast-feeding. In addition, a medically acceptable method of birth control must be used such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
7. Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms at least 30 days after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.
8. Subject agrees to refrain from taking multivitamins that include Ascorbic Acid and B-complex vitamins or a Magnesium supplement for a full 24 hours in advance of Week 1, Day 1 through the final Follow-up Visit, Day 174.

Clinical Exclusion Criteria

1. Inability to obtain informed consent.
2. Pregnancy or suspected pregnancy during study period. Subjects of childbearing potential must a have negative pregnancy test ≤ 7 days prior to treatment.
3. Recent diagnosis of cancer or treatment for cancer within last 12 months.
4. Life expectancy < 12 months.
5. CVA < 1 month prior to screening or any CVA resulting in unresolved walking impairment.
6. STEMI Myocardial infarction < 1 month prior to procedure.
7. Contraindication to contrast media or any study-required medication.
8. Coagulopathy or clotting disorders.
9. Suspected systemic infection affecting target limb.
10. Serum creatinine ≥ 2.5 mg/dL unless dialysis-dependent.
11. Enrollment in a drug study or medical device investigational research study.
12. Previous standard of care treatment to the same target lesion < 3 months prior to study enrollment.

Anatomic Exclusion Criteria

1. Greater than 50% DS following treatment of inflow lesions in the iliac or common femoral artery.
2. Unresolved complication following treatment of inflow lesions, or inflow lesion requiring a stent graft or surgical intervention.
3. Grade 4 or grade 5 stent fracture affecting target stent or proximal to the target stent.
4. Aneurysm within the target vessel.
5. Subjects with (or planned to receive) amputation(s) above the ankle, including major amputation, unilateral or bilateral.
6. Subject is expected to require further interventional standard of care treatment, during study participation (approximately 174 days).

Miscellaneous Exclusion Criteria

1. Standard of care cannot include drug eluting stent (DES).
2. Concurrent enrollment in another investigational drug or device study or has received other investigational drugs within 14 days of enrollment.
3. Had surgery within 4 weeks prior to study treatment except for the interventional standard of care.
4. Has a history of blood clots, pulmonary embolism, or deep vein thrombosis unless controlled by anticoagulant treatment.
5. Has a history of an arterial thromboembolic event within the prior six months including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina.
6. Has uncontrolled human immunodeficiency virus (HIV) infection or hepatitis B or C.
7. Has any clinically significant infection, i.e., any acute viral, bacterial, or fungal infection that requires specific treatment (anti-infective treatment has to be completed ≥ 7 days prior to study entry).
8. Has any other severe, uncontrolled medical condition, including uncontrolled diabetes mellitus (defined as a Hemoglobin A1C ≥ 9% in subjects with a prior history of diabetes, 28 days prior to study) or clinical signs of unstable congestive heart failure.
9. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
10. Prior allogeneic bone marrow or organ transplantation.
11. Grade 3 peripheral neuropathy within 14 days before enrollment.
12. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinical significant or baseline prolongation of the rate-corrected QT interval (e.g., repeated demonstration of QTc interval > 480 milliseconds).
13. Subject has other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or investigation product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for enrollment in this study.
14. Subject has any mental or medical condition that prevents the subject from giving informed consent or participating in the trial.
15. Subject has any condition that, in the opinion of the investigator, might jeopardize the safety of the subject or interfere with protocol compliance.
16. Prior history of sensitivity or allergic reaction to any of the following: Ascorbic Acid (Vitamin C), Magnesium Sulfate, Thiamine (b1), Cyanocobalamin (b12), Riboflavin (b2), Calcium D-Pantothenate (b5), Pyridoxine (b6), and Niacinamide (b3).

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Treatment-related Major Adverse Events as Defined by Re-intervention of the Target Vessel(s), Limb Amputation or Endovascular-related Death. | 84 days
  MAE rates compared to an objective performance criterion (historical control). MAEs are defined as re-intervention of the target vessel(s), amputation of all or part of the target limb, or endovascular-related death.

SECONDARY OUTCOMES:
Change of Walking Impairment Questionnaire Score Measured at Day 1 and Day 84 in Rejuveinix Treated Patients | 84 days
  Walking impairment questionnaire (WIQ), measured at Week 12, Day 84 (-2 to +14 days) compared to baseline assessed Week 1, Day 1 prior to administration of RJX.

IPD SHARING:
Plan to Share IPD: No